CLINICAL TRIAL: NCT01102816
Title: Acupuncture for Pain Management of Hemodialysis Patients: a Randomized, Controlled Pilot Study
Brief Title: Acupuncture for Pain Management of Hemodialysis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We failed to recruit enough patients by regular recruitment methods (i.e., newspaper ads, hospital postings, radios and television ads).
Sponsor: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Korea Institute of Oriental Medicine, Acupuncture, Moxibustion and Meridian Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KI0908; KI0908 (Other: Korea Institute of Oriental Medicine)
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: End-stage Renal Disease; Chronic Kidney Disease
Keywords: hemodialysis; end-stage renal disease; pain; acupuncture
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized acupuncture (Experimental)
  Interventions: Other: Individualized acupuncture treatment
- Routine care (No Intervention)
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Individualized acupuncture treatment — Individualized acupuncture treatment which focuses on each patient's symptoms and conditions will be provided twice a week for 6 weeks on a non-dialysis access day or before hemodialysis at dialysis-access day. 10-20 acupuncture needles will be inserted on the body except the arteriovenous fistula-located arm(s). Electrical stimulation of acupuncture will be conducted on 4 needles and the remained needles will be manipulated manually to elicit de-qi sensation. Needle retention time will be 20 minutes.
  Routine care provided by dialysis staffs, primary physicians and other healthcare providers will be maintained.
  Patients who received acupuncture treatment will be interviewed to explore patient's perceptions and experiences of acupuncture for their pain management. (Nested-qualitative study)
  Arms: Individualized acupuncture
Other: Routine care — Patients in this group will maintain routine care provided by their dialysis staffs, primary physicians or other healthcare providers for symptomatic care and disease management of end-stage renal disease through 6 weeks. After post-treatment evaluation, acupuncture treatment will be provided to patients who want to receive acupuncture treatment.
  Arms: Routine care

SUMMARY:
The purpose of this study is to determine the feasibility, effectiveness and safety of acupuncture for pain management in hemodialysis patients.

DETAILED DESCRIPTION:
Pain is one of the most common symptoms experienced by end-stage renal disease (ESRD) patients, which subsequently debilitates patient's quality of life. Although reducing pain is crucial to successful patient care in hemodialysis population, symptoms are often undertreated.Conventional pharmacological approaches are limited in dialysis population , given their altered pharmacokinetics and pharmacodynamic profiles and increased potential for adverse reactions. Acupuncture has been known to be beneficial in various chronic pain condition. As a non-pharmacologic intervention, it might be valuable for pain management in hemodialysis patients whose analgesic use are limited due to altered pharmacokinetics. However, little is known for the benefits of acupuncture for pain management in dialysis population. This study aims to determine whether acupuncture is a feasible, effective and safe therapeutic intervention for pain management in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* started hemodialysis at least 3 months ago
* receiving hemodialysis 3 times a week regularly
* equilibrated Kt/V ≥ 1.2
* pain occurred at least 3 months ago
* MYMOP2 symptom 1 score ≥ 3
* willingness to participate in this study

Exclusion Criteria:

* acute/chronic liver disease
* events of life-threatening cardiovascular disease within 6 months
* events of life-threatening neurological disorder within 6 months
* current/past history of neoplasm (in past 5 years)
* hemorrhagic disorder
* drug abuse/alcoholism
* other infectious disease
* history of the use of acupuncture, moxibustion or herbs within 1 month

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Pain measured on 0-6 scale of symptom 1 subscale score in the Measure Your Medical Outcome Profile2 (MYMOP2) questionnaire. | 6 weeks
  Patients will be asked to measure their pain on 0-6 scales (higher scores reflect worse pain) in the MYMOP2 questionnaire. Other subscales and summed profiles of MYMOP2 questionnaire will be regarded as secondary outcomes.

SECONDARY OUTCOMES:
Depressive moods measured by Beck Depression Inventory (BDI) | 6 weeks
  Follow-up evaluation will be conducted after 6 weeks from post-treatment measurement.
Quality of life of patients measured by Kidney Disease Quality of Life Version 1.3 (KDQOL-V 1.3) | 6 weeks
  Follow-up evaluation will be conducted after 6 weeks from post-treatment measurement.
Other patient-perceived changes on health and daily life measured by the MYMOP2 | 6 weeks
  Other changes of patients' health and daily life measured by Symptom 2(if measured), activity, and well-being subscales and total MYMOP2 profiles in the MYMOP2 questionnaire would be regarded as secondary outcomes. Follow-up evaluation will be conducted after 6 weeks from post-treatment measurememt.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Hyung Kim, MS, Principal Investigator — Korea Institute of Oriental Medicine
Locations (2):
- South Korea (2):
  - Korea Institute of Oriental Medicine (Clinical Research Center), Daejeon
  - Korea Institute of Oriental Medicine, Daejeon